CLINICAL TRIAL: NCT05691049
Title: Interventional, Post-marketing, Local, Mono-centric Study for Evaluation of Efficacy and Safety of HCC_45 for the Correction of Acne Scars of the Face
Brief Title: Evaluation of Efficacy and Safety of HCC_45 for the Correction of Acne Scars of the Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Collaborators: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0222
Record Dates: First submitted 2022-12-20; First posted 2023-01-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-01

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic; Ice Pick Scars; Rolling Scars; Boxcar Scars
Keywords: Acne scars; Hyaluronic acid; Ice pick Scars; Rolling scars; Boxcar scars
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Intervention Model Description: 30 subjects undergoing HCC_45 treatment of acne scars of the face by using a subcision + injection technique, the Needle (25 Gauge) or Cannula (25 Gauge) (wider areas are treated with Cannula) is inserted into the skin and made to move with a back-and-forth motion in order to detach scar collagen bundles. Then HCC_45 is injected. 3 visits: Day 0 (treatment) Day 30 (1 month after Day 0 treatment) Day 120 (4 months after Day 0 - follow-up).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCC_45 treatment group (Experimental): Treatment of acne scars of the face by using a subcision+injection technique: the needle (25 G) or cannula (25 G) (wider areas are treated with the cannula) is inserted into the skin and made to move with a back-and-forth motion in order to detach scar collagen bundles. Then 1 syringe (2 ml) of HCC_45 is injected.
  Day 0: Information and consent form provided, Clinical assessment, Digital clinical pictures, Instrumental assessment, Profilometry measurement.
  First treatment of HCC_45 (refer to study protocol).
  Day 30 (1 month after day 0): Clinical assessment, Digital clinical pictures, Instrumental assessment, Profilometry measurement.
  Second treatment of HCC_45 (refer to study protocol).
  Day 120 (4 months after day 0): Clinical assessment, Digital clinical pictures, Instrumental assessment, Profilometry measurement.
  NO treatment, Self-evaluation questionnaire.
  Interventions: Device: HCC_45

INTERVENTIONS:
Device: HCC_45 — Dosage form: HCC_45 is a resorbable medical device 2 ml non-pyrogenic pre-filled syringe, containing 2 ml of hyaluronic acid for intradermal use.
  The principal component of the medical device is Hyaluronic Acid of non-animal origin, produced by bacterial fermentation.

SUMMARY:
Acne scars represent a frequent complication of moderate/severe acne and may negatively impact on psychosocial and physical well-being of acne patients. Several types of acne scars have been classified and the same patient is likely to have more than one type. Each type can be treated with varying degrees of success. The main acne scars are the following:

Atrophic or Depressed Scarring:

* Ice pick: An ice pick scar has a wide shaft that narrows down to the tip. It resembles a hole that's wide at the top and narrows to a point as it goes deeper into the skin. Such an indentation is common and one of the most challenging scars to heal. This scar is more frequent on forehead and upper cheeks, where skin is thinner.
* Rolling: These scars are typically found on the lower cheeks and jaw, where skin is thicker. The indents have sloping edges that makes the skin look uneven and wavy.
* Boxcar: Boxcar scars are indents that have sharper edges. Those edges go down deep into the skin. These scars are common on the lower checks and jaw.

DETAILED DESCRIPTION:
Open label clinical trial, conducted by 1 center under dermatological control.

Primary aim of the study is to evaluate the efficacy and the safety of the deep injection of HCC_45 in acne scars of the face (ice picks, rolling, boxcars).

Secondary endpoint is self-assessment questionnaire regarding treatment efficacy and tolerance.

HCC_45 is a resorbable medical device 2 ml nonpyrogenic pre-filled syringe, containing 2 ml of hyaluronic acid for intradermal use. The principal component of the medical device is Hyaluronic Acid of non-animal origin, produced by bacterial fermentation.

ELIGIBILITY:
Inclusion Criteria:

* caucasian subjects of both sexes;
* age >18years
* asking for acne scars treatment;
* presenting acne scars (ice picks, rollings, boxcars);
* available and able to return to the study site for the post-procedural follow-up examinations;
* agreeing to present at each study visit without make-up;
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products;
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the Informed consent form.

Exclusion Criteria:

* Dependent on the volunteers' characteristics:
* smokers;
* performing in the 6 month before the trial beginning HA injections, radiofrequency treatment, toxin treatment;
* contraindication or know allergy to the devices' components or to the treatment;
* participation in a similar study actually or during the previous 3 months
* known pregnancy
* occurrence of pregnancy during the study
* Dependent on a clinical condition: Dermatological disease:
* Dermatitis;
* presence of cutaneous disease on the tested area,different from those under study
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne).
* Dependent on a clinical condition: General disease:
* Diabetes, coagulation disorders, connective tissue disorders, lipodystrophy or other systemic disease;
* HIV and/or immunosuppressive disease;
* cancerous or precancerous lesions in the either right or left midface;
* severe allergies manifested by a history of anaphylaxis, or history or presence of severe multiple allergies;
* alcohol or drug abusers;
* Dependent on a pharmacological treatment:
* Anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with except of contraceptive or hormonal treatment starting more than 1 year ago);
* assumption of drugs able to influence the test results in the investigator opinion.

The use of other drugs, not mentioned above, can be authorized by the Investigator. The trade name, the dosage, the start and stop date of the therapy will be reported on Case Record Form (CRF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Skin Roughness and flaccidity at 30 days and at 120 days post-injection | Day 0, Day 30, Day 120
  Visual score from 1 (milder scarring) to 4 (severe scarring) (Goodman and Baron Grading Scale of Postacne Scarring)
Change from Baseline of Skin's surface Profilometry at 30 days and at 120 days post-injection | Day 0, Day 30, Day 120
  A measurement of the skin surface affected by acne scars is taken thanks to Primos compact portable device (GFMesstechnik); Primos software is able to measure skin principal profilometric parameters in vivo or on skin replicas, the software compares directly the different images obtained at the times foresee by the protocol.

SECONDARY OUTCOMES:
Efficacy questionnaire | Day 120
  Self assessment questionnaire regarding the efficacy of the study treatment on acne scars (score: very marked; marked; medium; light; absent;)
Treatment tolerance questionnaire | Day 120
  Self-assessment score: bad; poor; good; excellent

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, MD, Principal Investigator — DERMING S.r.l., Clinical Research and Bioengineering Institute
Locations (1):
- DERMING S.r.l., Clinical Research and Bioengineering Institute, Milan, Lombardy, Italy

REFERENCES:
- [Derived] Sparavigna A, Grimolizzi F, Cigni C, Lualdi R, Bellia G. Dual-Plane Treatment With Highly Concentrated Hybrid Cooperative Complexes of Hyaluronans for Facial Atrophic Acne Scars. Dermatol Surg. 2025 Feb 1;51(2):152-156. doi: 10.1097/DSS.0000000000004387. Epub 2024 Oct 4. PMID 39365190